CLINICAL TRIAL: NCT01171885
Title: Evaluation of the Postoperative Analgesic Efficacy of Bilateral Superficial Cervical Block for Thyroidectomy and Mini Incision Under General Balanced Anesthesia: a Randomized, Triple Masked, Placebo Controlled Trial.
Brief Title: Bilateral Superficial Cervical Block for Thyroidectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lifecenter Hospital (Other)
Collaborators: Federal University of Minas Gerais (Other)
Responsible Party: Carlos Leonardo Alves Boni, Lifecenter Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE-0003.0.419.419-0
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2009-05

CONDITIONS: Cervical Pain
Keywords: Superficial cervical block; Thyroidectomy; Pain
MeSH Terms: conditions — Neck Pain; Pain | interventions — Saline Solution; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Bilateral superficial cervical block.
  Interventions: Drug: 0.9% saline
- Ropivacaine 0.25% (Experimental): Bilateral superficial cervical block
  Interventions: Drug: Ropivacaine
- Ropivacaine 0.5% (Experimental): Bilateral superficial cervical block.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: 0.9% saline — 20 ml of 0.9% saline
  Arms: Placebo
Drug: Ropivacaine — 20 ml of Ropivacaine 0.25%.
  Arms: Ropivacaine 0.25%
Drug: Ropivacaine — 20 ml of Ropivacaine 0.5%.
  Arms: Ropivacaine 0.5%

SUMMARY:
The objective of this study is to compare the postoperative analgesia afforded by bilateral superficial cervical block using different concentrations of local anesthetic (ropivacaine) in patients undergoing total thyroidectomy for the mini-incision technique, performed by the same surgical team.

DETAILED DESCRIPTION:
In this study we will evaluate the efficacy of bilateral superficial cervical block associated with balanced general anesthesia with remifentanil as opioid of choice in preventing postoperative pain in patients who underwent total thyroidectomy with mini incision without neck dissection.A hundred and twenty patients ASA I - II will be assessed and allocated randomly (through a table of random numbers) into three groups for analgesia for post-operative:

Group 1: bilateral superficial cervical block with 20 ml of 0.9% saline (placebo); Group 2: bilateral superficial cervical block with 20 ml ropivacaine 0.25%; Group 3: bilateral superficial cervical block with 20 ml ropivacaine 0.5%.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* Agreed to participate in the study and sign the consent form
* ASA I-II
* Scheduled to undergo total thyroidectomy without neck dissection under general balanced anesthesia.

Exclusion Criteria:

* Clinical history or laboratory tests suggestive of bleeding disorder
* Mental or cognitive deficit in existence, which makes it impossible to understand the patient visual analog scale of pain or the study protocol
* Body mass index greater than 45
* History of allergy to local anesthetics
* Intolerance or contraindication to any medication used in the study
* Skin infection at the site of the blockade
* Patients requiring neck dissection
* Pregnancy
* Preoperative use of opioid analgesics or non-opioids, corticosteroids or anti inflammatory non steroidal
* Patient's refusal to participate in the study
* Need for emergency reintervention within the first 24 hours postoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2009-07; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Post operative pain assessment according to Visual Analogue Scale | 24 Hours

SECONDARY OUTCOMES:
Consumption of morphine | 24 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Leonardo A Boni, MD, Principal Investigator — Federal University of Minas Gerais
Locations (1):
- Lifecenter Hospital, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- [Background] Andrieu G, Amrouni H, Robin E, Carnaille B, Wattier JM, Pattou F, Vallet B, Lebuffe G. Analgesic efficacy of bilateral superficial cervical plexus block administered before thyroid surgery under general anaesthesia. Br J Anaesth. 2007 Oct;99(4):561-6. doi: 10.1093/bja/aem230. Epub 2007 Aug 6. PMID 17681971
- [Background] Herbland A, Cantini O, Reynier P, Valat P, Jougon J, Arimone Y, Janvier G. The bilateral superficial cervical plexus block with 0.75% ropivacaine administered before or after surgery does not prevent postoperative pain after total thyroidectomy. Reg Anesth Pain Med. 2006 Jan-Feb;31(1):34-9. doi: 10.1016/j.rapm.2005.10.008. PMID 16418022
- [Background] Eti Z, Irmak P, Gulluoglu BM, Manukyan MN, Gogus FY. Does bilateral superficial cervical plexus block decrease analgesic requirement after thyroid surgery? Anesth Analg. 2006 Apr;102(4):1174-6. doi: 10.1213/01.ane.0000202383.51830.c4. PMID 16551919
- [Background] Steffen T, Warschkow R, Brandle M, Tarantino I, Clerici T. Randomized controlled trial of bilateral superficial cervical plexus block versus placebo in thyroid surgery. Br J Surg. 2010 Jul;97(7):1000-6. doi: 10.1002/bjs.7077. PMID 20632263